CLINICAL TRIAL: NCT03083184
Title: Evaluation of the Efficacy of an inTerdialytic "Ethanol 40% v/v - enoxapaRin 1000 U/mL" Lock solutioN to Prevent Tunnelled Catheter Infections in Chronic Hemodialysis Patients: a mulTi-centre, Randomized, Single Blind, Parallel Group studY (ETERNITY)
Brief Title: Evaluation of the Efficacy of an inTerdialytic "Ethanol 40% v/v - enoxapaRin 1000 U/mL" Lock solutioN to Prevent Tunnelled Catheter Infections in Chronic Hemodialysis Patients
Acronym: ETERNITY
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Ministry of Health, France (Other Government); CH du Puy en Velay, Hôpital Emile Roux (Unknown); University Hospital, Toulouse (Other); Centre hospitalier de Chambéry (Unknown); Calydial (Other); Hôpital Edouard Herriot (Other); Nouvel Hôpital Civil, 1 place de l'Hôpital 67091 Strasbourg cedex (Unknown); Hôpital Lapeyronie (Unknown); Centre de dialyse d'Alès (Unknown); University Hospital of Saint-Etienne (Other); Centre hospitalier de Perpignan (Other); Centre de néphrologie Polyclinique Médipôle Saint-Roch, Rue Ambroise Croizat (Unknown); CHU Hôpital Maison Blanche, 45 Rue Cognacq-Jay 51092 REIMS Cedex (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: CHU-0307; 2016-A00180-51 (Other: 2016-A00180-51)
Record Dates: First submitted 2017-03-07; First posted 2017-03-17 (Actual); Last update posted 2023-12-08 (Actual); Status verified 2023-05

CONDITIONS: Tunnelled Hemodialysis Catheter Infection
Keywords: Hemodialysis; hemodiafiltration; tunnelled dialysis catheter; interdialytic lock solution; preventing tunnelled catheter infection
MeSH Terms: interventions — Ethanol; Enoxaparin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Enrolled patients will be randomly assigned in a 1:1 ratio either to the intervention group (Ethenox) or to the control group (reference solution: UFH 5000 U/mL or citrate 4% w/v depending on which solution is generally used).
  Interventions: Drug: Ethanol
- control group (Other): Enrolled patients will be randomly assigned in a 1:1 ratio either to the intervention group (Ethenox) or to the control group (reference solution: UFH 5000 U/mL or citrate 4% w/v depending on which solution is generally used).
  Interventions: Drug: enoxaparin

INTERVENTIONS:
Drug: Ethanol — An ethanol 40 % v/v - enoxaparin 1000 U/mL (Ethenox) interdialytic lock solution
  Arms: Intervention group
Drug: enoxaparin — An ethanol 40 % v/v - enoxaparin 1000 U/mL (Ethenox) interdialytic lock solution
  Arms: control group

SUMMARY:
The purpose of this study is to assessed the efficacy of a combined solution of ethanol (4%) and low molecular weight heparins LMWH in preventing tunnelled dialysis catheter infection in chronic hemodialysis patients

DETAILED DESCRIPTION:
In France, a central venous catheter is used in 20 to 30% of chronic hemodialysis patients as the vascular access device. In this patient population the recommended device is a tunnelled dialysis catheter (TC). TC-related infections (TCI) and TC dysfunctions are two major complications and are associated with increased antibiotic consumption, hospital stays, health costs and mortality. Strategies to prevent TCI should target endoluminal biofilm formation, which is the major cause of long-term catheter colonization.

Unfractionated heparin (UFH), 5000 U/mL, is the standard interdialytic lock solution for the prevention of TC thrombosis. A lower-UFH concentration (1000U/mL) is associated with similar catheter patency. However, UFH has no antibiofilm properties. Antibiotic locks decrease the rate of TCI including TC- related bloodstream infections (TCBSI) and exit-site infection (ESI). The widespread use of antibiotic lock solutions raises concerns, however, because of side effects and the risk for the development of antimicrobial-resistant microorganisms.

Ethanol is an inexpensive antiseptic agent with activity against a broad range of bacteria and fungi commonly involved in TCI. It acts by non-specific protein denaturation and thus is less likely to promote antimicrobial resistance. Ethanol concentration of 40% v/v is highly effective in eradicating biofilm and has no significant impact on the integrity of silicone and polyurethane TCs or on their mechanical properties. A small randomized controlled trial performed in chronic hemodialysis patients with TC suggests that once-weekly instillation of an interdialytic ethanol lock is effective in preventing TCBSI. However, ethanol has no anticoagulant properties and may induce TC dysfunctions when used alone.

Experimental data provide evidence that a combined solution of ethanol and injectable anticoagulant is a promising lock solution for preventing both TC infections and dysfunctions. UFH, at whatever concentration, cannot be mixed with ethanol 40% v/v because of precipitation. ERA-EDTA recommends using low molecular weight heparins (LMWHs) for blood circuit anticoagulation during dialysis sessions. Like UFH, LMWHs have no antibiofilm properties. In contrast, LMWHs can be mixed in ethanol 40% v/v with enoxaparin having the highest solubility, up to 1300 U/mL. Our group demonstrated that ethanol 40% v/v - enoxaparin 400 U/mL is stable, compatible with TC materials and exhibits antibiofilm and anticoagulant properties in vitro (patent). No clinical studies have previously assessed the efficacy of a combined solution of ethanol and LMWH in preventing TCI in chronic hemodialysis patients.

Screening Patients eligible to participate in the study will be identified by a clinical research assistant in each study centre at the beginning of the study and then weekly. Data recorded in the medical records will be used.

Enrolment Eligible patients, previously identified during the screening procedure, will be recruited during a routine hemodialysis session by an investigator from centres participating in this study Randomization Enrolled patients will be randomly assigned in a 1:1 ratio either to the intervention group (Ethenox) or to the control group (reference solution: UFH 5000 U/mL or citrate 4% w/v depending on which solution is generally used). Random allocation will be performed by minimization using a computer algorithm. Minimization strata will be the study centre, the incident or prevalent nature of the TC and in the prevalent group the existence or not of a previous infection of the TC in place.

Single blind procedure The study will be performed single blind for the patients and the analysts. The recognisable smell of ethanol and the need to prepare the Ethenox lock solution rule out blinding of the healthcare staff.

Treatment Study treatment (Ethenox in the intervention group or reference solutions in the control group: UFH 5000 U/mL or citrate 4% w/v according to usual practice) will be used by the hemodialysis nurse as TC lock solution after each hemodialysis session with all successive TCs used during the study.

All the centres participating in the study will use similar hygiene protocols for TC placement and maintenance in accordance with the guidelines drawn up by the Haute Autorité de Santé and the Société Française d'Hygiène Hospitalière. Audits will be conducted during the study to ensure compliance with guidelines.

Study assessments Bacteriological sampling will be performed in accordance with guidelines for TCI.

A monthly blood sample will be taken as part of the routine care given to the patients.

Data will be collected weekly in an electronic case report form (e-CRF) except endpoint data for adjudication and serious adverse events, which will be recorded continuously.

ELIGIBILITY:
Inclusion Criteria:

* end-stage renal disease
* chronic hemodialysis/hemodiafiltration at least three times a week
* functional TC inserted for at least two weeks
* Social security cover
* Written informed consent

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2018-02-09 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Time to first TC infection (TCI) | at 1 year
  TCI is a composite endpoint defined by the occurrence of at least one of the three following events:
  Definitive TC-related bloodstream infection (definitive TCBSI) or Probable TC-related bloodstream infection (probable TCBSI) or TC exit-site infection (ESI). TCI diagnosis and its type (definitive or probable TCBSI or ESI) will be assessed by an endpoint adjudication committee (EAC) according to predefined criteria

SECONDARY OUTCOMES:
Time to first definitive or probable TCBSI | at 1 year
  TCI prevention criteria
Time to first ESI | at 1 year
  TCI prevention criteria
Incidence rate of definitive or probable TCBSI | at 1 year
  TCI prevention criteria
Incidence rate of ESI | at 1 year
  TCI prevention criteria
prevalence of colonizations of removed TCs for each TC removed | at 1 year
Incidence rate of TC dysfunctions | at 1 year
Dialysis dose measured by the dialysis machine | at 1 year
time to TC removal | at 1 year
Time to first systemic antibiotic treatment for TCI | at 1 year
Total duration ( type of antibiotic treatment) | at 1 year
Time to first hospitalization for TCI | at 1 year
Total duration of hospital stays for TCI | at 1 year
Total number of TCs replaced during the study | at 1 year
Incidence rate of breaches in TC integrity (TC leakage or disruption) | at 1 year
Incidence rate of clinical adverse events related to ethanol exposure | at 1 year
  Incidence rate of clinical adverse events related to ethanol exposure (tiredness, ethanol taste, headaches, dizziness, nausea, light-headedness, and increase in serum aspartate aminotransferase, alanine aminotransferase, gamma-glutamyl transferase or alkaline phosphatase).
Incidence rate of type II heparin-induced thrombocytopenia. | at 1 year
Incidence rate of hemorrhages | at 1 year
  bleeding or suspected bleeding, qualified as major if associated with a decrease in hemoglobin levels of more than 2g/dL or the need to transfuse at least two units of red blood cells

CONTACTS AND LOCATIONS:
Overall Officials: Julien ANIORT, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France

REFERENCES:
- [Derived] Aniort J, Piraud A, Adda M, Perreira B, Bouiller M, Fourcade J, Guerraoui A, Kalbacher E, Krumel T, Moragues HL, Thibaudin D, Vela CG, Vernin G, Weclawiak H, Bernard L, Heng AE, Souweine B. Evaluation of the efficacy of an interdialytic "ethanol 40% v/v - enoxaparin 1000 U/mL" lock solution to prevent tunnelled catheter infections in chronic hemodialysis patients: a multi-centre, randomized, single blind, parallel group study. BMC Nephrol. 2019 Apr 30;20(1):149. doi: 10.1186/s12882-019-1338-6. PMID 31039759